CLINICAL TRIAL: NCT05524038
Title: Comparison Between the Analgesic Effects of Ultrasound-guided Unilateral Quadratus Lumborum Block (Lateral Approach) Versus Erector Spinae Plane Block in Patients Undergoing Unilateral Lower Abdominal Surgery
Brief Title: Comparison Between the Quadratus Lumborum Block ,Erector Spinae Plane Block in Lower Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Rana Ahmed Abdelghaffar, lecturer of anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D237
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-02

CONDITIONS: Lower Abdominal Surgery
Keywords: Quadratus Lumborum; Erecto Spinae plane
MeSH Terms: interventions — Bupivacaine; Ultrasonography; Dexamethasone

STUDY DESIGN:
Intervention Model Description: 1. (QL) QLB group
  2. (ESB) group
Who Masked: Participant, Care Provider
Masking Description: Randomization will be done by random sequence number generated by the computer kept in sealed envelopes. Those envelopes will be opened on the day of surgery when the patient is in the operating room and participant will receive either (QLB) or (ESPB) as per the envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (QL) group (Active Comparator): In (QL) group, (lateral Approach) :patient receive this block with 20 mg bupivacaine hydrochloride plus 4mg dexamethasone
  Interventions: Drug: Bupivacaine Hydrochloride; Device: Ultrasound device; Drug: Dexamethasone; Device: echogenic needle
- (ESB) group (Active Comparator): In (ESB) group, Erector Spinae Plane Block: patient receive this block with 20 mg bupivacaine hydrochloride plus 4mg dexamethasone
  Interventions: Drug: Bupivacaine Hydrochloride; Device: Ultrasound device; Drug: Dexamethasone; Device: echogenic needle

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 20mg of Bupivacaine hydrochloride as local anesthetic will be used in (QL) group and (ESB) group
  Other Names: Marcaine 0.25%
Device: Ultrasound device — high-frequency linear probe covered with sterile sheath Active Array L12-4 (8-13MHz) of an ultrasound machine (Philips clear vue350, Philips Healthcare, Andover MA01810, USA) for performing the blocks .
Drug: Dexamethasone — injection of 4mg dexamethasone in each block
  Other Names: Dexamethasone 4mg/ml
Device: echogenic needle — 22- gauge, 50 mm echogenic needle (Stimuplex D; B Braun, Germany) for performing the blocks .

SUMMARY:
the purpose of study is comparison between the analgesic effect of two techniques in adult lower abdominal surgeries

DETAILED DESCRIPTION:
the study will be performed from November 2021 to January 2023 at Fayoum University hospital after approval of the local institutional ethics committee and local institutional review board .A detailed informed consent will be signed by the eligible participants before recruitment and randomization.

Preoperative preparations and Premedication :•

Both groups will be assessed by history taking, careful examination ,and laboratory investigations like:

Complete blood count (CBC), coagulation profile:(prothrombin concentration(PC),Partial thromboplastin time(PTT),International Normalized Ratio(INR) ) , kidney function, liver function, ECG for patient >40 years old or indicated cases, specific investigations to each disease

.•the investigators will teach the patients Visual Analogue Score (VAS) and train them.

Intra operative technique and management:

When patients reach Theater, standard American Society of Anesthesiology(ASA) monitoring by (noninvasive blood pressure (NIBP), pulse oximetry, electrocardiography, and capnography) will be applied.

the investigators will allocate basal data for each patient like: heart rate (HR), systolic and diastolic blood pressure, mean arterial blood pressure and arterial oxygen saturation will be recorded. Intravenous cannulation (IV) and intravenous fluid will be started. Intravenous Midazolam 0.03-0.05 mg/kg will be administered to all patients as premedication, Then the patients undergoing general anesthesia, At the first pre-oxygenation with O2100% for at least 3-5 min then the investigators will start Induction of anesthesia for both groups, general anesthesia will be induced with intravenous injection of fentanyl (1-2 µg/kg) and propofol (1, 5 - 2 mg/kg), and then atracurium (0.5 mg/kg) will be injected for endotracheal intubation. Mechanical ventilation will be maintained by controlled mechanical ventilation (CMV) mode with tidal volume ( 6-8ml /kg) with oxygen and air (50:50) with target of EtCo2≈ 30-40 mmHg, anesthesia will be maintained with isoflurane 1%-2% , Incremental dose of atracurium (0.1 mg/kg) will be given every 20 min or when needed. In addition, 0.5μg/kg fentanyl will be given intraoperatively once needed (increase of heart rate or NIBP more than 20% of the basal records) After endotracheal intubation and finishing the operation before awakening of patients the anesthesiologist will perform either the (QL) block technique or the (ESPB) block technique.

Statistical analysis:

The collected data will be organized, tabulated and statistically analyzed using SPSS software statistical computer package version 22 (SPSS Inc, USA). For quantitative data, the mean and standard deviation (SD) or median and interquartile range will be calculated. Independent-t test or Mann-Whitney U test, when appropriate, will be used as a test of significance. Qualitative data will be presented as number and percentages, chi square (χ2) will be used as a test of significance. For interpretation of results of tests of significance, significance will be adopted at P ≤ 0.05.

Sample size was calculated using (G power version 3). Minimal sample size of patients was 20 in each group needed to get power level 0.90, alpha level 0.05 (two tailed) and effect size of 1.08 for the overall dose of morphine. To overcome problem of loss of follow up, calculated sample size was increased by 20% to reach 24 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-60 years old.
* Patients scheduled for elective abdominal surgeries
* ASA classification I, II.
* Ability to sign the consent.

Exclusion Criteria:

* Patient refusal.
* Coagulation disorders.
* Skin lesions or infection at site of proposed needle.
* Known allergy to local anesthetics, or opioids.
* Patients suffering from neurological or mental disease.
* Opioid consumption 48 hours before the operation.
* Sever Obesity body mass index(BMI) >35
* Difficulty in Ultrasonographic identification.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours after the end of operation
  Millie gram

SECONDARY OUTCOMES:
Ease of performance. | during performance of the block
  time required to perform the block in minutes .
Bowel injury | 24hours after operation
  yes or no
intra vascular injection | 24hours after operation
  yes or no
Hematoma formation | 24hours after operation
  yes or no
Pruritus | 24hours after operation
  yes or no
Nausea | 24hours after operation
  yes or no
vomiting | 24hours after operation
  yes or no
patient satisfaction | 24 hours after operation
  According to a satisfaction score (poor = zero; fair = one; good = two; excellent= 3).

OTHER OUTCOMES:
time of first using of analgesic | 24 hours
  The time of first use of morphine in hours
Visual Analogue Score immediately . | 1 minute post operative
  measuring post operative pain level using Visual Analogue Score (VAS) range from (0) no pain to (10) sever pain immediately post operatively
Visual Analogue Score at (4) | 4 hour post operative
  measuring post operative pain level using Visual Analogue Score (VAS)at(4)hours post operatively
Visual Analogue Score at (8) | 8 hours post operative
  measuring post operative pain level using Visual Analogue Score (VAS)at(8)hours post operatively
Visual Analogue Score at (12) | 12 hours post operative
  measuring post operative pain level using Visual Analogue Score at(VAS)(12)hours post operatively
Visual Analogue Score at ( 24) | 24 hours post operative
  measuring post operative pain level using Visual Analogue Score (VAS)at(24)hours post operatively
Age | 1 hour before operation
  in years
Weight | 1 hour before operation
  in kg
height | 1 hour before operation
  meter
BMI | 1 hour before operation
  kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: rana A. Abdelghaffar, MD, Principal Investigator — faculty of medicine ,Fayum university
Locations (1):
- Fayoum University hospital, Al Fayyum, Fayoum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] El-Boghdadly K, Pawa A. The erector spinae plane block: plane and simple. Anaesthesia. 2017 Apr;72(4):434-438. doi: 10.1111/anae.13830. Epub 2017 Feb 11. No abstract available. PMID 28188611